CLINICAL TRIAL: NCT00347100
Title: Treatment of Early Insulinization With Glargine in Type 2 Diabetes Patients Uncontrolled on Sulfonylurea or Metformin Monotherapy
Brief Title: Insulin Glargine in Type 2 Diabetic Patients
Acronym: TARGET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_L_01051
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Glyburide; Gliclazide; Glipizide; Metformin

ARMS (2):
- 1 (Experimental): Administration of Insulin Glargine and Sulfonylurea or Metformin
  Interventions: Drug: Insulin Glargine; Drug: Metformin
- 2 (Active Comparator): Administration of Sulfonylurea or Metformin + a second Oral Anti Diabetic (OAD) among Glyburide, Glyclazide,Glimiperide,Glipizide or Metformin
  Interventions: Drug: Glyburide; Drug: Glyclazide; Drug: Glimiperide; Drug: Glipizide; Drug: Metformin

INTERVENTIONS:
Drug: Insulin Glargine — Throughout study period
  Arms: 1
Drug: Glyburide — Combination throughout the study period. Titrate to FPG ≤ 100 mg/dl.
  Arms: 2
Drug: Glyclazide — Combination throughout the study period. Titrate to FPG ≤ 100 mg/dl.
  Arms: 2
Drug: Glimiperide — Combination throughout the study period. Titrate to FPG ≤ 100 mg/dl.
  Arms: 2
Drug: Glipizide — Combination throughout the study period. Titrate to FPG ≤ 100 mg/dl.
  Arms: 2
Drug: Metformin — Combination throughout the study period. Titrate to FPG ≤ 100 mg/dl.

SUMMARY:
Primary:

* To investigate the efficacy of insulin glargine (in terms of change in A1c from baseline to endpoint A1c < 7%)

Secondary:

* To investigate the safety of insulin glargine (in terms of hypoglycaemia, including symptomatic, non-symptomatic and nocturnal hypoglycaemia)
* To investigate whether beta cell function is preserved if this therapy is initiated before 2nd OAD (oral anti-diabetic drug) failure

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients with first OAD (Sulfonylurea [SU] or Metformin) failure
* Patients who are insulin naive (unless it was used for gestational diabetes or if insulin therapy was less than 1 week)
* Serum creatinine ≤ 1.5mg/dL
* BMI: 21-41 kg/m²
* 7.5%< A1c <11%
* Fasting plasma glucose > 7.5mmol/L
* On diet and exercise therapy and stable OAD treatment (SU or metformin > ½ maximal dose)for more than 1 month prior to enrolment
* Women not of childbearing potential (sterilization procedure done or menopausal > 2 years), or if of childbearing potential, agree to take reliable contraceptive measures during the study
* Able and willing to monitor blood glucose
* Able and willing to perform 7 point blood glucose self monitoring at baseline, 12 week and 24 week
* Understand that there is a 50% chance of being randomized to the insulin treatment arm and is willing to self inject insulin

Exclusion Criteria:

* Type 1 diabetes
* Acute complication of diabetes, such as diabetic ketoacidosis and hyperosmolar coma
* Pregnancy, breast-feeding
* People who work night shifts
* Hypersensitivity to investigational drugs or its additives, or intolerability to metformin
* Need for use of medications prohibited by the protocol during the study for treatment purpose
* Significant diseases in cardiovascular, liver, nerve, endocrine or other systems, unable to complete the study or difficult to be used in study analysis
* Drugs or alcohol abuse

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
A1c values | At baseline and 24 weeks

SECONDARY OUTCOMES:
Adverse events including hypoglycemia | From the beginning to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Jolain, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Beijing, China